CLINICAL TRIAL: NCT01791205
Title: A Multi-Center Observational Study on the Use of Biologic Drugs as Monotherapy or Combination With DMARDs in Patients With Rheumatoid Arthritis in Italian Clinical Practice (ARMONIA)
Brief Title: ARMONIA: An Observational Study of Biologic Drugs in Monotherapy or Combination With DMARDs in Italian Clinical Practice and the Efficacy and Safety of RoActemra/Actemra (Tocilizumab) Monotherapy in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28552
Record Dates: First submitted 2013-02-12; First posted 2013-02-13 (Estimated); Results first posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (2):
- Monotherapy: Eligible participants who received any biologic drug as a monotherapy in the 12 months prior to the study entry will be observed for Phase I. Participants who were enrolled in Phase I and received tocilizumab (TCZ) as a monotherapy will be observed for 18 months from the first infusion of TCZ in Phase II, where TCZ was prescribed according to the approved product information, local treatment guidelines and/or routine clinical practice.
- Combination Therapy: Eligible participants who received any biologic drug in combination with disease-modifying anti-rheumatic drugs (DMARDs) in the 12 months prior to study entry will be observed for Phase I.

SUMMARY:
This is a multicenter observational study in patients with rheumatoid arthritis in routine clinical practice in Italy. In the retrospective Part 1 of the study, clinical and demographic factors associated with the use of a biologic drug in monotherapy as compared to therapy in combination with Disease-modifying anti-rheumatic drugs (DMARDs) will be evaluated. In the retrospective/prospective Part 2 of the study, efficacy and safety of the use of RoActemra/Actemra (tocilizumab) in monotherapy will be evaluated. Patients will be followed for up to18 months.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* Adult patients, >/= 18 years of age
* Diagnosis of rheumatoid arthritis according to American College of Rheumatology (ACR)/ European League Against Rheumatism (EULAR) criteria
* Patients who received at least one cycle of biologic therapy, either in monotherapy or in combination, in the 12 months preceding the opening of the first site

Part 2:

* Patients on monotherapy with RoActemra/Actemra already enrolled in Part 1 of the study

Exclusion Criteria:

* Patients simultaneously participating in other studies with RoActemra/Actemra at the time of signing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis who have received at least one cycle of therapy with a biologic drug in monotherapy or in combination with DMARDs
Sampling Method: Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- Italy (23):
  - Bari, Apulia
  - Martina Franca, Apulia
  - Reggio Calabria, Calabria
  - Napoli, Campania
  - Telese Terme, Campania
  - Bologna, Emilia-Romagna
  - Rome, Lazio
  - Legnano, Lombardy
  - Milan, Lombardy
  - Monza, Lombardy
  - Pavia, Lombardy
  - Turin, Piedmont
  - Sassari, Sardinia
  - Ancona, The Marches
  - Iesi, The Marches
  - Florence, Tuscany
  - Pisa, Tuscany
  - Prato, Tuscany
  - Siena, Tuscany
  - Perugia, Umbria
  - Cona (Ferrara), Veneto
  - Padua, Veneto
  - Verona, Veneto

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 304 participants were enrolled in the study conducted from May 2013 to October 2014 at 29 centers in Italy.
Groups:
- Monotherapy: Eligible participants who received any biologic drug as a monotherapy in the 12 months prior to the study entry were observed for Phase I. Participants who were enrolled in Phase I and received tocilizumab (TCZ) as a monotherapy were observed for 18 months from the first infusion of TCZ in Phase II, where TCZ was prescribed according to the approved product information, local treatment guidelines and/or routine clinical practice.
- Combination Therapy: Eligible participants who received any biologic drug in combination with disease-modifying anti-rheumatic drugs (DMARDs) in the 12 months prior to study entry were observed for Phase I.
Period: Phase I
Arm/Group | Monotherapy | Combination Therapy
Started | 152 | 152
Completed | 152 | 152
Not Completed | 0 | 0
Period: Phase II
Arm/Group | Monotherapy | Combination Therapy
Started | 104 (Participants who received tocilizumab monotherapy in Phase I was observed in Phase II.) | 0
Completed | 92 | 0
Not Completed | 12 | 0
Not completed — Lack of Efficacy | 6 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Safety | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Remission of disease | 1 | 0
Not completed — Physician's decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all enrolled participants.
Groups:
- Monotherapy: Eligible participants who received any biologic drug as a monotherapy in the 12 months prior to the study entry were observed for Phase I. Participants who were enrolled in Phase I and received TCZ as a monotherapy were observed for 18 months from the first infusion of TCZ in Phase II, where TCZ was prescribed according to the approved product information, local treatment guidelines and/or routine clinical practice.
- Total: Total of all reporting groups
Arm/Group | Monotherapy | Combination Therapy | Total
Number analyzed (Participants) | 152 | 152 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (12.5) | 59.4 (10.9) | 58.4 (11.8)
Gender [Count of Participants; unit: Participants]
  Female | 130 | 127 | 257
  Male | 22 | 25 | 47

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Participants With Demographic Characteristics in Monotherapy and Combination Therapy
Description: Demographic characteristics were analyzed in participants at Baseline, where Baseline is considered as the study entry visit (day of informed consent form signed). Demographic characteristics which were taken into account included age in years, race, height in centimeters (cm), weight in Kilograms (Kg), and Body Mass Index (BMI) in Kg/cm^2. Participants with age =<, > 59 years, height =<, > 163 cm, weight =<, > 65.85 Kg and BMI =<, > 24.98 Kg/cm^2 are reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants. Participants with available data at specified time points are denoted as 'n'.
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 152 | 152
Participants
  Age =< 59 years (n= 152, 152) | 79 | 75
  Age > 59 years (n= 152, 152) | 73 | 77
  Race Caucasian (n= 152, 152) | 152 | 150
  Height =< 163 cm (n= 149, 150) | 81 | 69
  Height >163 cm (n= 149, 150) | 68 | 81
  Weight =< 65.85 Kg (n= 152, 152) | 84 | 68
  Weight > 65.85 Kg, (n= 152, 152) | 68 | 84
  BMI =< 24.98 Kg/cm^2 (n= 149, 150) | 77 | 74
  BMI > 24.98 Kg/cm^2 (n= 149, 150) | 72 | 76

2. Primary Outcome: Phase I: Number of Participants With Disease Duration in Monotherapy and Combination Therapy
Description: The duration of disease is defined as the total time from the diagnosis of rheumatoid arthritis (RA) until the study entry.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 152 | 152
Participants
  Duration of disease =< 124 months | 74 | 81
  Duration of disease > 124 months | 78 | 71

3. Primary Outcome: Phase I: Number of Participants With Comorbidity in Monotherapy and Combination Therapy
Description: Comorbidity is the presence of previous or concomitant diseases.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 152 | 152
Participants | 121 | 116

4. Primary Outcome: Phase I: Number of Participants With Autoantibody Status (Rheumatoid Factor and Anti-cyclic Citrullinated Protein Antibodies) in Monotherapy and Combination Therapy
Description: The autoantibody included seropositive or seronegative participants for rheumatoid factor (RF) and/or anti-cyclic citrullinated protein antibodies (Anti-CCP). RF value higher than 20 Units (U)/milliliter (mL) is considered seropositive and anti-CCP antibodies value higher than 10 U/mL is considered positive.
Time Frame: At Baseline (Day of informed consent form signed)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 128 | 128
Participants
  RF Positive (n= 128, 128) | 69 | 79
  RF Negative (n= 128, 128) | 59 | 49
  Anti-CCP Positive (n= 100, 103) | 61 | 72
  Anti-CCP Negative (n= 100, 103) | 39 | 31

5. Primary Outcome: Phase I: Number of Participants With Health Assessment Questionnaire- Disability Index in Monotherapy and Combination Therapy
Description: The Health Assessment Questionnaire- Disability Index (HAQ-DI) is a participant-reported questionnaire that measured quality of life in terms of physical function of participants with rheumatoid arthritis. It consisted of 20 questions in eight domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities) rated on a 4-point scale, where 0 (equals) = without difficulties; 1= with some difficulties; 2= with great difficulties; and 3= unable to perform these actions at all. The HAQ-DI scale was an average of all the scores and ranged from 0 (mild disability) to 3 (severe disability), where higher scores represents higher disease activity. Participants assessed their ability to do each task over the past seven days. Participants with scores =< 0.8625 and > 0.8625 are reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants. Participants with available data at the time of evaluation are reported.
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 84 | 80
Participants
  HAQ-DI Score =< 0.8625 | 42 | 40
  HAQ-DI Score >0.8625 | 42 | 40

6. Primary Outcome: Phase I: Number of Participants With Disease Activity Score 28 in Monotherapy and Combination Therapy
Description: The disease activity included Disease Activity Score 28 (DAS28). The DAS28 is a combined index for measuring disease activity in RA. The index includes swollen joint counts (SJC) and tender joint counts (TJC), acute phase response, and general health status. The DAS28 scale ranges from 0 to 10 (0= no disease activity and 10= maximum disease activity; where higher scores represents higher disease activity. The DAS =< 2.8 indicates clinical remission, >2.8 to 10 = low disease activity, >10 to 22 = moderate disease activity, and >22 = high disease activity. Participants with DAS28 score =< 2.6 and > 2.6 are reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants. Participants with available data at Baseline are reported.
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 121 | 122
Participants
  DAS28 with =< 2.6 score | 67 | 55
  DAS28 with >2.6 score | 54 | 67

7. Primary Outcome: Phase I: Number of Participants With C-Reactive Protein Value and Erythrocyte Sedimentation Rate in Monotherapy and Combination Therapy
Description: The disease activity included biological markers of inflammation: C-Reactive Protein (CRP) and Erythrocyte Sedimentation Rate (ESR). A reduction in CRP and ESR values indicates improvement. Participants with CRP values =< 0.28 and >2.8 milligram/deciliter (mg/dL); and ESR values =< 11 and >11 millimeters/hour (mm/hr) are reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants. Participants with available data at Baseline are reported. Participants with available data at specified time points are denoted as 'n'.
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 135 | 136
Participants
  CRP =< 0.28 mg/dL (n= 128, 129) | 66 | 64
  CRP > 0.28 mg/dL (n= 128, 129) | 62 | 65
  ESR =< 11 mm/h (n= 135, 136) | 80 | 59
  ESR > 11 mm/h (n= 135, 136) | 55 | 77

8. Primary Outcome: Phase I: Number of Participants With Clinical Disease Activity Index in Monotherapy and Combination Therapy
Description: The disease activity included Clinical Disease Activity Index (CDAI) which is the numerical sum of four outcome parameters: TJC and SJC based on a 28-joint assessment; and patient's global assessment (PtGA) and physician's global assessment (PhGA) assessed on 0-10 cm visual analog scale (VAS), where 0 = no disease activity and 10 = worst disease activity, where higher scores represents higher disease activity. The CDAI total score ranges from 0 (no disease activity) to 76 (maximal disease activity), where higher scores represents higher disease activity. The CDAI =< 2.8 indicates clinical remission, > 2.8 to 10 indicates low disease activity, > 10 to 22 indicates moderate disease activity, and > 22 indicates high disease activity. Participants with CDAI score =< 7.75 and > 7.75 are reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants. Participants with available data at Baseline are reported.
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 74 | 77
Participants
  CDAI Score =< 7.75 | 37 | 39
  CDAI Score > 7.75 | 37 | 38

9. Primary Outcome: Phase I: Number of Participants With Simplified Disease Activity Index in Monotherapy and Combination Therapy
Description: The disease activity included Simplified Disease Activity Index (SDAI) which is the numerical sum of five outcome parameters: TJC and SJC (based on a 28-joint assessment), PtGA and PhGA (based on 0-10 cm VAS, where 0 = no disease activity and 10 = worst disease activity), and CRP. SDAI total score ranges from 0 (no disease activity) to 86 (maximal disease activity), where higher scores represents higher disease activity. The SDAI =< 3.3 indicates disease remission, > 3.4 to 11 indicates low disease activity, > 11 to 26 indicates moderate disease activity, and > 26 indicates high disease activity. Participants with SDAI score =< 8.17 and > 8.17 are reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants. Participants with available data at Baseline are reported.
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 72 | 69
Participants
  SDAI Score =< 8.17 | 36 | 35
  SDAI Score > 8.17 | 36 | 34

10. Primary Outcome: Phase I: Number of Participants With Duration of Combination Therapy Before Monotherapy in Monotherapy and Combination Therapy
Description: The duration of combination therapy before monotherapy are reported. The duration was estimated by calculating total duration from starting the combination therapy till the participant switched to monotherapy. Participants who started the combination therapy and later switched to monotherapy =< 337 days, > 337 days, =< 336 days, > 336 days are reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 81 | 74
Participants
  Duration of combination type 1, =< 337 (n= 81, 74) | 45 | 33
  Duration of combination type 1, > 337 (n= 81, 74) | 36 | 41
  Duration of combination type 2, =< 336 (n= 64, 60) | 36 | 26
  Duration of combination type 2, > 336 (n= 64, 60 ) | 28 | 34

11. Primary Outcome: Phase I: Number of Participants Treatment Line in Which Monotherapy Has Been Adopted in Monotherapy
Description: The first biologic treatment line was defined as the first use of any biologic drug in treatment of rheumatoid arthritis, regardless its association with DMARDs and the second treatment line as the subsequent use of a different biologic drug. Participants who adopted monotherapy as =< 2 and > 2 therapy lines are reported. According to the study protocol objectives, this analysis was performed only for Monotherapy arm.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Monotherapy
Number analyzed (Participants) | 152
Participants
  Treatment line, =< 2 | 106
  Treatment line, > 2 | 46

12. Primary Outcome: Phase I: Number of Biologics Administered as Monotherapy in Monotherapy and Combination Therapy
Description: Participants who received at least one previous treatment with biologics in monotherapy and no previous monotherapy with biologics are reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 152 | 152
Participants
  No biologics | 95 | 125
  At least one biologics | 57 | 27

13. Primary Outcome: Phase I: Number of Participants With Prevalence of Previous Therapy Switches and Swaps in Monotherapy and Combination Therapy
Description: Participants who had prevalence with at least one previous switch, swaps, and switch/swap to other therapy are reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 152 | 152
Participants
  At least one switch | 30 | 40
  At least one swap | 74 | 56
  At least one switch/swap | 81 | 75

14. Primary Outcome: Phase I: Number of Participants With Reasons Leading to the Use of Biologic in Monotherapy
Description: Reasons leading to the use of biologic in monotherapy includes DMARDs intolerance, insufficient therapeutic effect, intolerance to biologic drug, low participant's compliance, concomitant pathologies, pregnancy desire, remission from combination therapy, remission from monotherapy, others and unknown. Participants with reason leading to the use of biologic in monotherapy are presented. According to the study protocol objectives, this analysis was performed only for Monotherapy arm.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Monotherapy
Number analyzed (Participants) | 152
Participants
  DMARDs intolerance | 41
  Insufficient therapeutic effect | 68
  Intolerance to biologic drug | 7
  Low participant compliance | 5
  Concomitant pathologies | 4
  Pregnancy desire | 3
  Remission from combination therapy | 9
  Remission from monotherapy | 3
  Others | 8
  Unknown | 3

15. Primary Outcome: Phase II: Percentage of Participants Who Retained on Tocilizumab Monotherapy
Description: The probabilities of participant to retain on therapy at various time points are reported.
Time Frame: Up to 18 months
Population: Analysis population included participants who were enrolled in Phase I and received tocilizumab as monotherapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Monotherapy
Number analyzed (Participants) | 104
Percentage of participants
  Day 1 | 99.0 [93.4 to 99.9]
  Day 33 | 97.1 [91.3 to 99.1]
  Day 66 | 96.2 [90.1 to 98.5]
  Day 168 | 95.2 [88.8 to 98.0]
  Day 236 | 94.2 [87.6 to 97.4]
  Day 323 | 93.3 [86.4 to 96.7]
  Day 375 | 92.3 [85.2 to 96.1]
  Day 414 | 91.3 [84.0 to 95.4]
  Day 423 | 90.4 [82.9 to 94.7]
  Day 442 | 89.4 [81.7 to 94.0]
  Day 459 | 88.5 [80.6 to 93.3]

16. Primary Outcome: Phase II: Retention Rate in Therapy, Percentage of Participants Achieving DAS 28 ESR <2.6 and <3.2 at Month 18
Description: Participants who retained the therapy were analyzed for disease activity (DAS28 ESR) at Month 18. The DAS28 ESR is a measure of the participant's disease activity calculated using TJC (28 joints), SJC (28 joints), PtGA using 0-10 cm VAS (0 = no disease activity and 10 = worst disease activity), and ESR. It is calculated by using the following formula: DAS28 ESR = 0.56 x square root of TJC + 0.28 x square root of SJC + 0.70 x log n at ESR + 0.014 x PtGA. The DAS28 ESR scores ranged from 0.49 (less disease activity) to 9.07 (maximal disease activity); decrease in score indicated improvement of disease.
Time Frame: At month 18
Population: Analysis population included participants who were enrolled in Phase I and received tocilizumab as monotherapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Monotherapy
Number analyzed (Participants) | 104
Percentage of participants
  DAS28 ESR<2.6 | 64.71 [51.13 to 78.28]
  DAS 28 ESR > 2.6 to =<3.2 | 80.39 [69.11 to 91.67]
Statistical Analysis 1: Comparison: Monotherapy; The relation between retention rate and DAS28 (<2.6 vs <3.2) was assayed with the Cox regression; Test type: Superiority or Other; p = 0.1194, Regression, Cox — The relation between retention rate and duration of disease for phase II was estimated with the Cox regression model; Hazard Ratio (HR) = 3.538, 95% CI 2-sided [0.65 to 19.33]

17. Secondary Outcome: Phase I: Median Disease Duration in Monotherapy and Combination Therapy
Description: The duration of disease is defined as the total time from the diagnosis of RA until the study entry.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Combination Therapy: Eligible participants who received any biologic drug in combination with DMARDs in the 12 months prior to study entry were observed for Phase I.
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 152 | 152
Months | 125 [111 to 150] | 114 [98 to 133]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.3895, Regression, Cox

18. Secondary Outcome: Phase I: Percentage of Participants With Comorbidity in Monotherapy and Combination Therapy
Description: Comorbidity is the presence of previous or concomitant diseases. Percentage of participants with comorbidity is reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 152 | 152
Percentage of participants | 79.61 | 76.32
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.4900, Regression, Logistic; Odds Ratio (OR) = 1.211, 95% CI 2-sided [0.703 to 2.086]

19. Secondary Outcome: Phase I: Mean Health Assessment Questionnaire-Disability Index in Monotherapy and Combination Therapy
Description: The HAQ-DI is a participant-reported questionnaire that measured quality of life in terms of physical function of participants with rheumatoid arthritis. It consisted of 20 questions in eight domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities) rated on a 4-point scale, where 0 (equals) = without difficulties; 1= with some difficulties; 2= with great difficulties; and 3= unable to perform these actions at all. The HAQ-DI scale was an average of all the scores and ranged from 0 (mild disability) to 3 (severe disability), where higher scores represents higher disease activity. Participants assessed their ability to do each task over the past seven days.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants.
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 152 | 152
Scores on scale | 0.873 (0.686) | 0.915 (0.667)
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.6908, t-test, 2 sided; Delta = -0.042, 95% CI 2-sided [-0.251 to 0.167]

20. Secondary Outcome: Phase I: Percentage of Participants Who Started Treatment With a Biologic Drug in Monotherapy and Percentage of Participants Who Stopped a DMARDs While Taking a Biologic Drug in Combination Therapy
Description: The table below shows percentage participants who started treatment with a biologic drug in monotherapy compared with percentage of participants who stopped DMARDs while taking a biologic drug in combination.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants. One participant in monotherapy group and 4 participants in combination group were not included because they had not received a previous treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 151 | 148
Percentage of Participants | 49.01 [40.9 to 57.1] | 35.81 [28.0 to 43.6]
Statistical Analysis 1: Comparison: Monotherapy vs Combination Therapy; Test type: Superiority or Other; p = 0.0210, Pearson's chi-squared test

21. Secondary Outcome: Phase I: Number of Participants Receiving a Biologic Drug as Monotherapy at Different Treatment Lines
Description: The first biologic treatment line was defined as the first use of any biologic drug in treatment of rheumatoid arthritis, regardless its association with DMARDs, the second treatment line as the subsequent use of a different biologic drug and so on for the third, fourth, fifth and sixth treatment line. According to the study protocol objectives, this analysis was performed only for Monotherapy arm.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants.
Measure: Number; unit: Participants
Arm/Group | Monotherapy
Number analyzed (Participants) | 152
Participants
  Treatment Line 1 | 71
  Treatment Line 2 | 35
  Treatment Line 3 | 35
  Treatment Line 4 | 6
  Treatment Line 5 | 4
  Treatment Line 6 | 1

22. Secondary Outcome: Phase I: Number of Participants With at Least One Previous Treatment With Biologics Drug as a Monotherapy in Monotherapy and Combination Therapy
Description: Number of participants who received at least one previous treatment with a biologic drug as a monotherapy in both groups is reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: as for outcome 20
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 151 | 148
Participants | 57 | 27

23. Secondary Outcome: Phase I: Percentage of Participants With Prevalence of Previous Therapy Switches and Swaps in Monotherapy and Combination Therapy
Description: Participants who had prevalence with at least one previous switch, swaps or switch/swap to other therapy either monotherapy or combination therapy are reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 152 | 152
Percentage of participants
  Switch | 19.74 [13.34 to 26.14] | 26.32 [19.24 to 33.40]
  Swap | 48.68 [40.65 to 56.72] | 36.84 [29.09 to 44.60]
  Switch/Swap | 53.29 [45.27 to 61.31] | 49.34 [41.30 to 57.38]

24. Secondary Outcome: Phase I: Median DAS28 at Study Entry in Monotherapy and Combination Therapy
Description: The DAS28 is a combined index for measuring disease activity in RA. The index includes SJC and TJC, acute phase response, and general health status. The DAS28 scale ranges from 0 to 10 (0= no disease activity and 10= maximum disease activity) where higher scores represents higher disease. The DAS28 <2.6 indicates disease remission, >=2.6 and <3.2 indicates Low disease activity, >=3.2 and <=5.1 indicates Moderate disease activity and >5.1 indicates High disease activity. Median score for DAS28 at the study entry (Baseline) is reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants. Participants with available DAS28 score at Baseline are reported.
Measure: Median (Full Range); unit: Scores on scale
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 121 | 122
Scores on scale | 2.51 [0.77 to 6.28] | 2.77 [0.28 to 6.27]

25. Secondary Outcome: Phase I: Number of Participants With CDAI Scores at Study Entry in Monotherapy and Combination Therapy
Description: The CDAI is the numerical sum of four outcome parameters: TJC and SJC based on a 28-joint assessment; and PtGA and PhGA assessed on 0-10 cm VAS, where 0 = no disease activity and 10 = worst disease activity, where higher scores represents higher disease activity. The CDAI total score ranges from 0 (no disease activity) to 76 (maximal disease activity), where higher scores represents higher disease activity. The CDAI =< 2.8 indicates clinical remission, > 2.8 to 10 indicates low disease activity, > 10 to 22 indicates moderate disease activity, and > 22 indicates high disease activity. Number of participants with CDAI scores for both the groups at study entry (baseline) are reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants. Participants with available CDAI score at Baseline are reported.
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 74 | 77
Participants
  Disease remission | 18 | 16
  Low disease activity | 28 | 30
  Moderate disease activity | 20 | 21
  High disease activity | 8 | 10

26. Secondary Outcome: Phase I: Number of Participants With SDAI Scores at Study Entry in Monotherapy and Combination Therapy
Description: The SDAI is the numerical sum of five outcome parameters: TJC and SJC (based on a 28-joint assessment), PtGA and PhGA (assessed on 0-10 cm) VAS; 0 = no disease activity and 10 = worst disease activity), and CRP (mg/dL). SDAI total score ranges from 0 (no disease activity) to 86 (maximal disease activity), where higher scores represents higher disease activity. The SDAI =< 3.3 indicates disease remission, > 3.4 to 11 indicates low disease activity, > 11 to 26 indicates moderate disease activity, and > 26 indicates high disease activity.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants. Participants with available SDAI score at Baseline are reported.
Measure: Number; unit: Participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 72 | 69
Participants
  Disease remission | 19 | 17
  Low disease activity | 25 | 26
  Moderate disease activity | 22 | 20
  High disease activity | 6 | 6

27. Secondary Outcome: Phase I: Mean Tender Joints and Swollen Joints as Disease Activity at Study Entry in Monotherapy and Combination Therapy
Description: Mean of tender and swollen joints was determined by examining 28 joints and identified the joints that were painful under pressure or to passive motion. The number of tender and swollen joints was recorded on the joint assessment as no tenderness = 0 and tenderness = 1.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants. Participants with available tender and swollen joints at Baseline are reported.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 138 | 133
Joints
  Tender Joints | 2.49 (3.30) | 2.71 (3.75)
  Swollen Joints | 1.29 (2.34) | 1.20 (2.45)

28. Secondary Outcome: Phase I: Percentage of Participants Treated With Corticosteroids at Study Entry in Monotherapy and Combination Therapy
Description: The percentage of participants treated with corticosteroids at enrollment is reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 152 | 152
Percentage of participants | 46.05 [38.04 to 54.07] | 55.26 [47.27 to 63.26]

29. Secondary Outcome: Phase I: Mean Dose of Corticosteroids At Study Entry in Monotherapy and Combination Therapy
Description: Mean dose of corticosteroids at study entry (Baseline) is reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants. Participants who received corticosteroids were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 70 | 84
milligrams | 4.64 (3.00) | 4.71 (3.12)

30. Secondary Outcome: Phase I: Mean Duration of Previous Treatment With a Biologic Drug in Monotherapy and Combination Therapy
Description: Mean duration of previous treatment with a biologic drug in monotherapy are reported.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants. Participants who received previous treatment with a biologic drug before monotherapy were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 46 | 22
Days | 1254.7 (816.0) | 1188.3 (995.0)

31. Secondary Outcome: Phase I: Mean Duration of Treatment With A Biologic Drug in Combination With DMARDs Before Monotherapy
Description: Mean duration of treatment with a biologic drug in combination with DMARDs before monotherapy is reported in days.
Time Frame: At Baseline (Day of informed consent form signed)
Population: Analysis population included all enrolled participants. Participants who received previous treatment with a biologic drug in combination with DMARDs before monotherapy were considered for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Monotherapy | Combination Therapy
Number analyzed (Participants) | 82 | 75
Days | 1486.1 (988.4) | 1525.9 (1132.1)

32. Secondary Outcome: Phase II: Percentage of Participants Maintaining Delta DAS 28 CRP of >= 0.6 at Months 3, 6, 12, and 18
Description: Participants who maintained the change in DAS28 (Delta DAS28) CRP of >=0.6 after 3, 6, 12, and 18 months from the first infusion with tocilizumab as monotherapy are reported. The DAS28-CRP is a combined index that measured RA disease activity. It is calculated using TJC (28 joints), SJC (28 joints), PtGA using 0-10 cm VAS (0 = no disease activity and 10 = worst disease activity), and CRP (mg/dL). It is calculated by using the formula: DAS28 CRP= 0.56 × square root of TJC 28 + 0.28 square root of SJC 28 + 0.36 × log n at (CRP+1) + 0.014 × PtGA + 0.96. The DAS28 CRP- scores ranged from 0.49 (less disease activity) to 9.07 (maximal disease activity); decrease in score indicated improvement of disease.
Time Frame: At Months 3, 6, 12, and 18
Population: Analysis population included participants who were enrolled in Phase I and received tocilizumab as monotherapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Monotherapy
Number analyzed (Participants) | 104
Percentage of participants
  Month 3 | 55.36 [41.92 to 68.79]
  Month 6 | 56.6 [42.81 to 70.4]
  Month 12 | 60.78 [46.92 to 74.65]
  Month 18 | 60 [45.94 to 74.06]

33. Secondary Outcome: Phase II: Percentage of Participants Maintaining Delta DAS28 ESR >= 0.6 at Months 3, 6, 12, and 18
Description: Participants who maintained delta DAS28 ESR of >= 0.6 after 3, 6, 12, and 18 months from the first infusion with tocilizumab as monotherapy are reported. The DAS28 ESR is a measure of the participant's disease activity calculated using TJC (28 joints), SJC (28 joints), PtGA using 0-10 cm VAS (0 = no disease activity and 10 = worst disease activity), and ESR. It is calculated by using the following formula: DAS28 ESR = 0.56 x square root of TJC + 0.28 x square root of SJC + 0.70 x log n at ESR + 0.014 x PtGA. The DAS28 ESR scores ranged from 0.49 (less disease activity) to 9.07 (maximal disease activity); where decrease in score indicated improvement of disease.
Time Frame: At Months 3, 6, 12, and 18
Population: Analysis population included participants who were enrolled in Phase I and received tocilizumab as monotherapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Monotherapy
Number analyzed (Participants) | 104
Percentage of participants
  Month 3 | 55.00 [42.04 to 67.96]
  Month 6 | 67.86 [55.24 to 80.48]
  Month 12 | 58.82 [44.84 to 72.8]
  Month 18 | 72.55 [59.87 to 85.23]

34. Secondary Outcome: Phase II: Percentage of Participants Achieving DAS28 CRP Remission (< 2.6) and Low Disease Activity (<3.2) at Months 3, 6, 12, and 18
Description: The DAS28-CRP is a combined index that measured RA disease activity. It is calculated using TJC (28 joints), SJC (28 joints), PtGA using 0-10 cm VAS (0 = no disease activity and 10 = worst disease activity), and CRP (mg/dL). It is calculated by using the formula: DAS28 CRP= 0.56 × square root of TJC (28 joints) + 0.28 square root of SJC (28 joints) + 0.36 × log n at (CRP+1) + 0.014 × PtGA + 0.96. The DAS28 CRP scores ranged from 0.49 (less disease activity) to 9.07 (maximal disease activity); decrease in score indicated improvement of disease. The DAS28 CRP < 2.6 indicates disease remission and >=2.6 to 3.2 indicates low disease activity.
Time Frame: At Months 3, 6, 12, and 18
Population: Analysis population included participants who were enrolled in Phase I and received tocilizumab as monotherapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Monotherapy
Number analyzed (Participants) | 104
Percentage of participants
  DAS28 CRP < 2.6, Month 3 | 18.18 [7.66 to 28.7]
  DAS28 CRP < 2.6, Month 6 | 43.1 [29.97 to 56.24]
  DAS28 CRP < 2.6, Month 12 | 64.15 [50.81 to 77.5]
  DAS28 CRP < 2.6, Month 18 | 60.78 [46.92 to 74.65]
  DAS28 CRP < 3.2, Month 3 | 32.73 [19.93 to 45.53]
  DAS28 CRP < 3.2, Month 6 | 67.24 [54.79 to 79.69]
  DAS28 CRP < 3.2, Month 12 | 84.91 [74.94 to 94.87]
  DAS28 CRP < 3.2, Month 18 | 76.47 [64.42 to 88.52]

35. Secondary Outcome: Phase II: Percentage of Participants Achieving DAS 28 ESR (< 2.6) and Low Disease Activity (<3.2) at Months 3, 6, 12, and 18
Description: The DAS28 ESR is a measure of the participant's disease activity calculated using TJC (28 joints), SJC (28 joints), PtGA using 0-10 cm VAS (0 = no disease activity and 10 = worst disease activity), and ESR. It is calculated by using the following formula: DAS28 ESR = 0.56 x square root of TJC + 0.28 x square root of SJC + 0.70 x log n at ESR + 0.014 x PtGA. The DAS28 ESR scores ranged from 0.49 (less disease activity) to 9.07 (maximal disease activity); decrease in score indicated improvement of disease. The DAS28 ESR < 2.6 indicates disease remission and >=2.6 to 3.2 indicates low disease activity.
Time Frame: At Months 3, 6, 12, and 18
Population: Analysis population included participants who were enrolled in Phase I and received tocilizumab as monotherapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Monotherapy
Number analyzed (Participants) | 104
Percentage of participants
  DAS28 ESR < 2.6, Month 3 | 14.04 [4.74 to 23.33]
  DAS28 ESR < 2.6, Month 6 | 42.62 [29.85 to 55.39]
  DAS28 ESR < 2.6, Month 12 | 53.57 [40.09 to 67.05]
  DAS28 ESR < 2.6, Month 18 | 64.71 [51.13 to 78.28]
  DAS28 ESR < 3.2, Month 3 | 24.56 [13.04 to 36.08]
  DAS28 ESR < 3.2, Month 6 | 70.49 [58.71 to 82.27]
  DAS28 ESR < 3.2, Month 12 | 83.93 [74.00 to 93.85]
  DAS28 ESR < 3.2, Month 18 | 80.39 [69.11 to 91.67]

36. Secondary Outcome: Phase II: Percentage of Participants Achieving CDAI Remission (< 2.8) at Months 3, 6, 12, and 18
Description: Percentage of participants achieving CDAI remission < 2.8, after 3, 6, 12 and 18 months from the first infusion with tocilizumab as monotherapy are reported. CDAI is the numerical sum of four outcome parameters: TJC, SJC based on a 28-joint assessment; and PtGA and PhGA assessed on 0-10 cm VAS, where 0 = no disease activity and 10 = worst disease activity, where higher scores represents higher disease activity. The CDAI total score ranges from 0 (no disease activity) to 76 (maximal disease activity), where higher scores represents higher disease activity. The CDAI =< 2.8 indicates clinical remission, > 2.8 to 10 indicates low disease activity, > 10 to 22 indicates moderate disease activity, and > 22 indicates high disease activity.
Time Frame: At Months 3, 6, 12, and 18
Population: Analysis population included participants who were enrolled in Phase I and received tocilizumab as monotherapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Monotherapy
Number analyzed (Participants) | 104
Percentage of participants
  Month 3 | 11.11 [0.33 to 21.9]
  Month 6 | 16.67 [3.88 to 29.46]
  Month 12 | 33.33 [17.16 to 49.51]
  Month 18 | 31.58 [16.1 to 47.06]

37. Secondary Outcome: Phase II: Percentage of Participant Achieving SDAI Remission (< 3.3) at Months 3, 6, 12, and 18
Description: Percentage of participant achieving SDAI remission (< 3.3), after 3, 6, 12 and 18 months from the first infusion with tocilizumab as monotherapy is reported. The SDAI is the numerical sum of five outcome parameters: TJC and SJC (based on a 28-joint assessment), PtGA and PhGA which (based on 0-10 cm VAS, 0 = no disease activity and 10 = worst disease activity, where higher scores represent higher disease activity), and CRP. The SDAI total score ranges from 0 (no disease activity) to 86 (maximal disease activity), where higher scores represents higher disease activity. The SDAI =< 3.3 indicates disease remission, > 3.4 to 11 = low disease activity, > 11 to 26 = moderate disease activity, and > 26 = high disease activity.
Time Frame: At Months 3, 6, 12, and 18
Population: Analysis population included participants who were enrolled in Phase I and received tocilizumab as monotherapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Monotherapy
Number analyzed (Participants) | 104
Percentage of participants
  Month 3 | 12.5 [0.39 to 24.61]
  Month 6 | 22.22 [7.96 to 36.49]
  Month 12 | 50.00 [32.29 to 67.71]
  Month 18 | 36.36 [19.04 to 53.69]

38. Secondary Outcome: Phase II: Mean Change From Baseline in TJC And SJC at Months 3, 6, 12, and 18
Description: The mean change from Baseline (day of the first infusion with tocilizumab as monotherapy) in the TJC And SJC after 3, 6, 12 and 18 months is reported. The TJC and SJC were determined for 28 joint counts. The scores ranged from 0 (no disease activity) to 28 (higher/worsen disease activity), where higher scores represents higher disease activity.
Time Frame: From Baseline (Day of first administration of TCZ as a monotherapy) to Months 3, 6, 12, and 18
Population: Analysis population included participants who were enrolled in Phase I and received tocilizumab as monotherapy. Participants with available data at specified time points are denoted as 'n'.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Monotherapy
Number analyzed (Participants) | 80
Joints
  TJC, Month 3 (n= 78) | -2.74 (6.87)
  TJC, Month 6 (n= 80) | -4.13 (5.51)
  TJC, Month 12 (n= 72) | -4.33 (6.14)
  TJC, Month 18 (n= 69) | -4.30 (5.89)
  SJC, Month 3 (n= 78) | -1.65 (3.98)
  SJC, Month 6 (n= 80) | -2.39 (3.47)
  SJC, Month 12 (n= 72) | -2.21 (3.76)
  SJC, Month 18 (n= 69) | -2.46 (3.75)

39. Secondary Outcome: Phase II: Mean Change From Baseline in Dose of Corticosteroids at Months 3, 6, 12, and 18
Description: Mean Change From Baseline (day of the first infusion with tocilizumab as monotherapy) in the dose of corticosteroids after 3, 6, 12 and 18 months from Baseline is reported.
Time Frame: From Baseline (Day of first administration of TCZ as a monotherapy) to Months 3, 6, 12, and 18
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Monotherapy
Number analyzed (Participants) | 60
milligrams
  Month 3 (n= 60) | -0.85 (4.18)
  Month 6 (n= 54) | -1.24 (2.28)
  Month 12 (n= 41) | -1.71 (2.76)
  Month 18 (n= 38) | -1.08 (2.12)

40. Secondary Outcome: Phase II: Percentage of Participants With Delta HAQ >= 0.21 at Months 3, 6, 12, and 18
Description: Percentage of participants with change in HAQ (Delta HAQ) of >= 0.21 after 3, 6, 12 and 18 months from the first infusion with tocilizumab as monotherapy are reported. The HAQ consisted of 20 questions in eight domains (dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities) rated on a 4-point scale, where 0 (equals) = without difficulties; 1= with some difficulties; 2= with great difficulties; and 3= unable to perform these actions at all. The HAQ-DI scale was an average of all the scores and ranged from 0 (mild disability) to 3 (severe disability), where higher scores represents higher disease activity.
Time Frame: At Months 3, 6, 12, and 18
Population: Analysis population included participants who were enrolled in Phase I and received tocilizumab as monotherapy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Monotherapy
Number analyzed (Participants) | 104
Percentage of participants
  Month 3 | 8.51 [0.23 to 16.79]
  Month 6 | 10.00 [0.28 to 19.72]
  Month 12 | 13.89 [2.02 to 25.76]
  Month 18 | 8.11 [0.00 to 17.33]

41. Secondary Outcome: Phase II: Mean VAS Fatigue Score Overtime
Description: The VAS fatigue score ranging from 0 (symptom-free and no arthritis symptoms) to 100 (worsening in symptoms and arthritis disease activity). Higher score indicate worsening.
Time Frame: At Baseline (Day of first administration of TCZ as a monotherapy) and Months 3, 6, 12, and 18
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Monotherapy
Number analyzed (Participants) | 24
Scores on scale
  Baseline (n= 19) | 54.95 (25.49)
  Month 3 (n= 24) | 40.58 (20.67)
  Month 6 (n= 24) | 30.42 (21.20)
  Month 12 (n= 17) | 33.82 (23.72)
  Month 18 (n= 23) | 23.35 (25.01)

42. Secondary Outcome: Phase II: Number of Participants With Any Adverse Events, Any Serious Adverse Events, Adverse Events of Special Interest, and Tubercular Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable or unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Pre-existing conditions that worsened during the study were reported as AE. A serious adverse event (SAE) is any untoward medical occurrence that at any dose results in death is life threatening, requires hospitalization or prolongation of hospitalization, or results in disability/incapacity, or congenital anomaly/birth defect. The AE were captured only for Phase II.
Time Frame: Up to 18 months
Population: Analysis population included participants who were enrolled in Phase I and received tocilizumab as monotherapy.
Measure: Number; unit: Participants
Arm/Group | Monotherapy
Number analyzed (Participants) | 104
Participants
  Any AE | 56
  Any SAE | 5
  AE/SAE of special interest | 10
  Tubercular AE/SAE | 0

43. Secondary Outcome: Phase II: Number of Participants With Retention in Therapy Without Interruption Due to Side Effects
Description: Number of participants who retained in therapy without interruption due to side effects is reported.
Time Frame: Up to 18 months
Population: Analysis population included participants who were enrolled in Phase I and received tocilizumab as monotherapy.
Measure: Number; unit: Participants
Arm/Group | Monotherapy
Number analyzed (Participants) | 104
Participants | 103

44. Secondary Outcome: Phase II: Number of Side Effects That Had Not Induced Discontinuation of Treatment
Description: Number of side effects (AEs) that had not induced discontinuation of treatment is reported. The AEs were captured only for Phase II.
Time Frame: Up to 18 months
Population: Analysis population included participants who were enrolled in Phase I and received tocilizumab as monotherapy.
Measure: Number; unit: AEs
Arm/Group | Monotherapy
Number analyzed (Participants) | 104
AEs | 19

45. Secondary Outcome: Phase II: Number of Side Effects That Induced Transient Interruption of Treatment
Description: Number of side effects (AEs) that induced transient interruption of treatment is reported. The AEs were captured only for Phase II.
Time Frame: Up to 18 months
Population: Analysis population included participants who were enrolled in Phase I and received tocilizumab as monotherapy.
Measure: Number; unit: AEs
Arm/Group | Monotherapy
Number analyzed (Participants) | 104
AEs | 15

46. Secondary Outcome: Phase II: Mean Change From Baseline in Hemoglobin Levels Over Time
Description: The mean change in hemoglobin concentration was calculated by subtracting the baseline hemoglobin concentration from the monthly hemoglobin concentration is reported.
Time Frame: From Baseline (Day of first administration of TCZ as a monotherapy) to Months 3, 6, 12, and 18
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: gram/dL
Arm/Group | Monotherapy
Number analyzed (Participants) | 84
gram/dL
  Month 3 (n= 83) | 0.41 (0.84)
  Month 6 (n= 84) | 0.34 (0.91)
  Month 12 (n= 80) | 0.44 (1.01)
  Month 18 (n= 76) | 0.49 (1.16)

47. Secondary Outcome: Phase II: Mean Change From Baseline in Hematocrit, Neutrophils, Eosinophils, Basophils, Lymphocytes, and Monocytes Over Time
Description: Mean Change from Baseline in hematocrit, neutrophils, eosinophils, basophils, lymphocytes, monocytes are reported.
Time Frame: From Baseline (Day of first administration of TCZ as a monotherapy) to Months 3, 6, 12, and 18
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Percentage of cells
Arm/Group | Monotherapy
Number analyzed (Participants) | 64
Percentage of cells
  Hematocrit, Month 3 (n= 60) | 5.73 (36.25)
  Hematocrit, Month 6 (n= 57) | -0.11 (7.12)
  Hematocrit, Month 12 (n= 57) | 0.32 (7.26)
  Hematocrit, Month 18 (n= 53) | -0.35 (8.35)
  Neutrophils, Month 3 (n= 61) | -7.82 (11.96)
  Neutrophils, Month 6 (n= 64) | -7.69 (11.35)
  Neutrophils, Month 12 (n= 57) | -7.16 (11.99)
  Neutrophils, Month 18 (n= 55) | -6.69 (13.32)
  Eosinophils, Month 3 (n= 58) | 1.21 (2.54)
  Eosinophils, Month 6 (n= 59) | 1.25 (2.11)
  Eosinophils, Month 12 (n= 52) | 1.30 (2.49)
  Eosinophils, Month 18 (n= 51) | 1.31 (2.16)
  Basophils, Month 3 (n= 58) | 0.14 (0.67)
  Basophils, Month 6 (n= 59) | 0.26 (0.63)
  Basophils, Month 12 (n= 52) | 0.19 (0.47)
  Basophils, Month 18 (n= 51) | 0.18 (0.41)
  Lymphocytes, Month 3 (n= 60) | 5.58 (9.05)
  Lymphocytes, Month 6 (n= 64) | 5.60 (9.50)
  Lymphocytes, Month 12 (n= 57) | 4.98 (9.67)
  Lymphocytes, Month 18 (n= 55) | 4.55 (11.45)
  Monocytes, Month 3 (n= 58) | 0.61 (2.87)
  Monocytes, Month 6 (n= 59) | 1.13 (2.75)
  Monocytes, Month 12 (n= 52) | 0.46 (2.38)
  Monocytes, Month 18 (n= 51) | 0.59 (2.74)

48. Secondary Outcome: Phase II: Mean Change From Baseline in Red Blood Cells, White Blood Cells, and Platelets Over Time
Description: Mean change from baseline in red blood cells (RBC), white blood cells (WBC) and platelets are reported.
Time Frame: From Baseline (Day of first administration of TCZ as a monotherapy) to Months 3, 6, 12, and 18
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: 10^6 cells/microliter
Arm/Group | Monotherapy
Number analyzed (Participants) | 84
10^6 cells/microliter
  RBC, Month 3 (n= 71) | 0.07 (0.32)
  RBC, Month 6 (n= 70) | -0.01 (0.30)
  RBC, Month 12 (n= 69) | 0.04 (0.32)
  RBC, Month 18 (n= 63) | 0.05 (0.29)
  WBC, Month 3 (n= 83) | -1.14 (2.01)
  WBC, Month 6 (n= 84) | -1.30 (2.27)
  WBC, Month 12 (n= 81) | -1.30 (2.09)
  WBC, Month 18 (n= 75) | -1.48 (2.15)
  Platelets, Month 3 (n= 78) | -52.38 (71.21)
  Platelets, Month 6 (n= 75) | -62.12 (72.58)
  Platelets, Month 12 (n= 73) | -54.42 (73.40)
  Platelets, Month 18 (n= 72) | -57.88 (76.15)

49. Secondary Outcome: Phase II: Mean Change From Baseline in Total Cholesterol, Low-density and High-density Lipoprotein Cholesterol, Triglycerides, Total Bilirubin, Direct Bilirubin, Glucose, Creatinine, Blood Urea Nitrogen Levels Over Time
Description: Mean change from baseline in total cholesterol, low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, triglycerides (TG), total bilirubin, direct bilirubin, glucose, creatinine, blood urea nitrogen (BUN) levels are reported.
Time Frame: From Baseline (Day of first administration of TCZ as a monotherapy) to Months 3, 6, 12, and 18
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Monotherapy
Number analyzed (Participants) | 64
mg/dL
  Total Cholesterol, Month 3 (n= 27) | 10.04 (42.31)
  Total Cholesterol, Month 6 (n= 28) | 12.61 (49.76)
  Total Cholesterol, Month 12 (n= 31) | 4.81 (41.59)
  Total Cholesterol, Month 18 (n= 28) | 5.57 (49.00)
  LDL Cholesterol, Month 3 (n= 14) | -3.63 (24.89)
  LDL Cholesterol, Month 6 (n= 14) | 13.93 (38.99)
  LDL Cholesterol, Month 12 (n= 16) | -2.59 (37.10)
  LDL Cholesterol, Month 18 (n= 14) | 3.53 (38.31)
  HDL Cholesterol, Month 3 (n= 19) | 4.16 (6.34)
  HDL Cholesterol, Month 6 (n= 18) | 0.67 (11.42)
  HDL Cholesterol, Month 12 (n= 19) | -1.74 (12.61)
  HDL Cholesterol, Month 18 (n= 18) | -1.67 (15.46)
  TG, Month 3 (n= 23) | -7.91 (45.29)
  TG, Month 6 (n= 27) | -2.78 (50.39)
  TG, Month 12 (n= 26) | 2.85 (53.05)
  TG, Month 18 (n= 27) | 12.93 (71.09)
  Total Bilirubin, Month 3 (n= 5) | 0.28 (0.29)
  Total Bilirubin, Month 6 (n= 9) | 0.18 (0.45)
  Total Bilirubin, Month 12 (n= 9) | 0.04 (0.28)
  Total Bilirubin, Month 18 (n= 7) | 0.36 (0.74)
  Direct Bilirubin, Month 3 (n= 5) | 0.08 (0.17)
  Direct Bilirubin, Month 6 (n= 9) | 0.06 (0.28)
  Direct Bilirubin, Month 12 (n= 9) | 0.03 (0.28)
  Direct Bilirubin, Month 18 (n= 7) | 0.13 (0.21)
  Glucose, Month 3 (n= 16) | 2.50 (9.00)
  Glucose, Month 6 (n= 21) | 4.13 (29.90)
  Glucose, Month 12 (n= 24) | 8.24 (27.36)
  Glucose, Month 18 (n= 20) | -2.10 (26.15)
  Creatinine, Month 3 (n= 60) | -0.02 (0.20)
  Creatinine, Month 6 (n= 64) | -0.21 (1.29)
  Creatinine, Month 12 (n= 60) | -0.33 (1.60)
  Creatinine, Month 18 (n= 53) | -0.38 (1.70)
  BUN, Month 3 (n= 22) | 1.31 (8.87)
  BUN, Month 6 (n= 25) | 1.14 (8.80)
  BUN, Month 12 (n= 24) | -0.18 (8.31)
  BUN, Month 18 (n= 22) | 0.06 (8.91)

50. Secondary Outcome: Phase II: Mean Change From Baseline in Aspartate Transaminase, Alanine Transaminase, Gamma-glutamyl Transpeptidase, and Alkaline Phosphatase Levels Over Time
Description: Mean change from baseline in aspartate transaminase (AST), alanine transaminase (ALT), gamma-glutamyl transpeptidase (GGT) and alkaline phosphatase levels are reported.
Time Frame: From Baseline (Day of first administration of TCZ as a monotherapy) to Months 3, 6, 12, and 18
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Units/Liter
Arm/Group | Monotherapy
Number analyzed (Participants) | 76
Units/Liter
  AST, Month 3 (n= 74) | 0.75 (9.35)
  AST, Month 6 (n= 74) | 0.87 (9.39)
  AST, Month 12 (n= 74) | 0.78 (8.47)
  AST, Month 18 (n= 68) | 1.53 (13.40)
  ALT, Month 3 (n= 74) | 3.08 (20.65)
  ALT, Month 6 (n= 76) | 0.60 (20.49)
  ALT, Month 12 (n= 76) | 0.08 (16.15)
  ALT, Month 18 (n= 68) | 0.22 (18.27)
  GGT, Month 3 (n= 25) | -0.84 (20.45)
  GGT, Month 6 (n= 32) | -6.19 (24.68)
  GGT, Month 12 (n= 30) | -4.60 (21.50)
  GGT, Month 18 (n= 25) | -7.48 (26.50)
  Alkaline phosphatase, Month 3 (n= 20) | -15.10 (38.22)
  Alkaline phosphatase, Month 6 (n= 21) | -21.86 (38.02)
  Alkaline phosphatase, Month 12 (n= 24) | -18.17 (44.29)
  Alkaline phosphatase, Month 18 (n= 15) | -21.60 (53.45)

51. Secondary Outcome: Phase II: Mean Change From Baseline in Serum Electrophoresis Parameters Over Time
Description: Serum electrophoresis parameters includes albumin, alpha-1 globulin, alpha-2 globulin, beta globulin, gamma globulin was reported. Mean change from Baseline values are reported at each time points.
Time Frame: From Baseline (Day of first administration of TCZ as a monotherapy) to Months 3, 6, 12, and 18
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: Percentage of concentration
Arm/Group | Monotherapy
Number analyzed (Participants) | 26
Percentage of concentration
  Albumin, Month 3 (n= 25) | 3.92 (4.23)
  Albumin, Month 6 (n= 25) | 5.23 (3.29)
  Albumin, Month 12 (n= 24) | 5.35 (5.14)
  Albumin, Month 18 (n= 19) | 5.95 (4.45)
  Alpha-1 globulin, Month 3 (n= 26) | -0.85 (0.94)
  Alpha-1 globulin, Month 6 (n= 25) | -1.09 (0.91)
  Alpha-1 globulin, Month 12 (n= 25) | -1.00 (1.10)
  Alpha-1 globulin, Month 18 (n= 19) | -1.11 (1.03)
  Alpha-2 globulin, Month 3 (n= 25) | -1.74 (2.12)
  Alpha-2 globulin, Month 6 (n= 25) | -1.68 (2.30)
  Alpha-2 globulin, Month 12 (n= 24) | -1.91 (1.95)
  Alpha-2 globulin, Month 18 (n= 19) | -2.34 (1.89)
  Beta globulin, Month 3 (n= 25) | -0.94 (1.36)
  Beta globulin, Month 6 (n= 24) | -1.19 (1.43)
  Beta globulin, Month 12 (n= 24) | -0.91 (1.41)
  Beta globulin, Month 18 (n= 19) | -1.07 (1.18)
  Gamma globulin, Month 3 (n= 25) | -0.51 (1.96)
  Gamma globulin, Month 6 (n= 26) | -1.75 (3.46)
  Gamma globulin, Month 12 (n= 24) | -1.51 (2.44)
  Gamma globulin, Month 18 (n= 19) | -1.52 (2.62)

ADVERSE EVENTS:
Time Frame: Up to 18 months
Description: AEs are collected for participants who were enrolled in Phase I and received TCZ as a monotherapy for 18 months from the first infusion of TCZ in Phase II. AEs were not collected for participants who received Combination therapy.
Arm/Group | Monotherapy
Serious Adverse Events (participants affected / at risk) | 5/104
Other Adverse Events (participants affected / at risk) | 54/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy (N=104)
Otitis externa (Infections and infestations) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monotherapy (N=104)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Osteoporosis (Metabolism and nutrition disorders) | 1
Hypogammaglobulinaemia (Immune system disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Neutrophil count decreased (Investigations) | 1
Ultrasound kidney abnormal (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Hysteroscopy (Investigations) | 1
Transaminases increased (Investigations) | 1
Gengival abscess (Infections and infestations) | 1
Bacteriuria (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 5
Genital candidasis (Infections and infestations) | 1
Vulvovaginal candidasis (Infections and infestations) | 1
Keratitis viral (Infections and infestations) | 1
Cystitis (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Upper respiratory tract infection bacterial (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Wound infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiovascular disorder (Cardiac disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 8
Polycythaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Ligament sprain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Lumbar vertebral fracture (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Congenital neurological disorder (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 1
Keratitis (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 3
Otitis media (Ear and labyrinth disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Herpes zoster (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Tooth abscess (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Pharyngitis (Gastrointestinal disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Gastroenteritis viral (Gastrointestinal disorders) | 2
Oral herpes (Gastrointestinal disorders) | 1
Gastrointestinal infection (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Procedural vomiting (Gastrointestinal disorders) | 1
Cystitis bacterial (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Musculoskeletal chest pain (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Influenza (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Rinitis (Respiratory, thoracic and mediastinal disorders) | 2
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillitis streptococcal (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Influenza like illness (General disorders) | 1
Hypertensive crisis (Vascular disorders) | 3
Hypertension (Vascular disorders) | 2
Withdrawal hypertension (Vascular disorders) | 1
Essential hypertension (Vascular disorders) | 1
Syncope (Vascular disorders) | 1
Anal fistula excision (Surgical and medical procedures) | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 1
Dental operation (Surgical and medical procedures) | 1
Foot operation (Surgical and medical procedures) | 1
Uterine polypectomy (Surgical and medical procedures) | 1
Synovectomy (Surgical and medical procedures) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Wound infection (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights